CLINICAL TRIAL: NCT02477267
Title: A Pivotal, Phase 1, Open-Label, Randomized, Crossover, Single-Dose, Comparative Bioavailability Study of Buprenorphine-Naloxone Sublingual Spray and Suboxone® Sublingual Film in Healthy Volunteers
Brief Title: Study of Buprenorphine-Naloxone Sublingual Spray and Suboxone® Sublingual Film in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: INSYS Therapeutics Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: INS009-15-033
Record Dates: First submitted 2015-06-18; First posted 2015-06-22 (Estimated); Last update posted 2015-09-03 (Estimated); Status verified 2015-08

CONDITIONS: Opiate Dependence
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Buprenorphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test-Reference Sequence (Experimental): SL spray, followed by SL film
  Interventions: Drug: SL spray; Drug: SL film
- Reference-Test Sequence (Experimental): SL film followed by SL spray
  Interventions: Drug: SL spray; Drug: SL film

INTERVENTIONS:
Drug: SL spray
  Other Names: Buprenorphine naloxone sublingual spray
Drug: SL film
  Other Names: Buprenorphine and naloxone sublingual film

SUMMARY:
The primary objective of this study is to compare the bioavailability of a test formulation of Buprenorphine Naloxone Sublingual (SL) spray to that of a single dose of Suboxone® (buprenorphine and naloxone) sublingual film, under fasted conditions.

ELIGIBILITY:
Inclusion Criteria:

* Meets protocol-specified criteria for qualification and contraception
* Is willing and able to remain confined in the study unit for the entire duration of each treatment period and comply with restrictions related food, drink and medications
* Voluntarily consents to participate and provides written informed consent prior to any protocol-specific procedures

Exclusion Criteria:

* Has history or current use of over-the-counter medications, dietary supplements, or drugs (including nicotine and alcohol) outside protocol-specified parameters
* Has signs, symptoms or history of any condition that, per protocol or in the opinion of the investigator, might compromise:

  1. the safety or well-being of the participant or study staff;
  2. the safety or well-being of the participant's offspring (such as through pregnancy or breast-feeding);
  3. the analysis of results

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2015-06; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration (Cmax) | within 21 days
  Categories: buprenorphine, norbuprenorphine, unconjugated naloxone, and total naloxone
Time to Cmax (Tmax) | within 21 days
  Categories: buprenorphine, norbuprenorphine, unconjugated naloxone, and total naloxone
Elimination rate constant | within 21 days
  Categories: buprenorphine, norbuprenorphine, unconjugated naloxone, and total naloxone
Elimination half-life (T½) | within 21 days
  Categories: buprenorphine, norbuprenorphine, unconjugated naloxone, and total naloxone
Area under the curve to the final sample with a concentration greater than the limit of quantification (LOQ [AUClast]) | within 21 days
  Categories: buprenorphine, norbuprenorphine, unconjugated naloxone, and total naloxone
Area under the curve extrapolated to infinity (AUCinf) | within 21 days
  Categories: buprenorphine, norbuprenorphine, unconjugated naloxone, and total naloxone

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni DeCastro, Study Director — INSYS Therapeutics Inc
Locations (1):
- Worldwide Clinical Trials Early Phase Services, LLC, San Antonio, Texas, United States